CLINICAL TRIAL: NCT06780774
Title: Investigating the Acute and Chronic Effects of a Supplement Containing Caffeine, Vitamins, Minerals and Botanical Extracts on Cognition, Sleep and Wellbeing, in Healthy Volunteers.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 67G1
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-11

CONDITIONS: Caffeine; Sleep; Cognitive Function; Wellbeing; Mood
Keywords: Caffeine; Cognitive function; Sleep; Wellbeing; Mood
MeSH Terms: interventions — Caffeine; Vitamins; Minerals

STUDY DESIGN:
Intervention Model Description: Randomised, double-blind, placebo-controlled, crossover design.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Treatment will be blinded according to the randomisation schedule by a researcher who has no other involvement in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Caffeine, Vitamins, Minerals and Botanical Blend (Capsule) (Experimental): Blend containing 120mg of caffeine, vitamins, minerals and botanical extracts in capsule form. The treatment will be consumed daily, for 29 days, as one bolus dose (2 capsules).
  Interventions: Dietary Supplement: Caffeine, Vitamins, Minerals and Botanical Blend
- Placebo (Capsule) (Placebo Comparator): Blend containing 17mg Marigold Extract and Brown rice flour, in capsule form. The treatment will be consumed daily, for 29 days, as one bolus dose (2 capsules).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Caffeine, Vitamins, Minerals and Botanical Blend — Blend containing 120mg of caffeine, vitamins, minerals and botanical extracts in capsule form.
  Other Names: Active Treatment
  Arms: Caffeine, Vitamins, Minerals and Botanical Blend (Capsule)
Dietary Supplement: Placebo — Blend containing 17mg Marigold Extract and Brown rice flour. Other Names: Placebo Treatment
  Arms: Placebo (Capsule)

SUMMARY:
The aim of the study is to investigate the acute and chronic effects of a supplement containing Caffeine, Vitamins, Minerals and Botanical extracts on cognitive function, sleep and wellbeing, in healthy volunteers.

The study will follow a randomised, double-blind, placebo-controlled, crossover design. Participants will receive both treatments, and both study arms will include an acute testing visit (day 1) and a chronic testing visit (day 29). The active treatment contains a blend of 120mg caffeine, vitamins, minerals and botanical extracts and the matched placebo treatment contains marigold extract and brown rice flour.

The trial will use computerised cognitive tasks, administered via COMPASS software (Northumbria University, UK), online cognitive assessments via Cognimapp and self-reported questionnaires and sleep diary, as measures of the outcome variables.

90 participants will participate, aged 18-75, and self-ported as being in good health. Participants will be randomly allocated to a treatment order and will be supplied with either the active treatment or the placebo whilst visiting the research centre for the acute testing visits. Participants will take the treatment home to consume daily for the duration of the supplementation period. Participants will record the time of taking treatment each day in a treatment diary which will be returned to the research centre, along with any unused treatment, at each chronic testing visit.

DETAILED DESCRIPTION:
The study will follow a randomised, placebo-controlled, double-blind, crossover design. Participants will first receive either the active treatment (a blend containing 120mg caffeine, vitamins, minerals and botanical extracts) or a matched placebo (containing 17mg Marigold extract and brown rice flour), for 29 days before crossing over to the other treatment condition for a further 29 days. Participants will attend all 6 appointments required, 5 of which will be at the research centre, will complete at home treatment diary daily, as well as completing the at home assessments.

Participants will initially attend a virtual screening appointment (conducted via telephone call or Microsoft Teams) which will involve obtaining informed consent, health screening, completion of the Caffeine Consumption Questionnaire (CCQ) and collection of demographic information. Participants will then attend the research centre on five occasions.

The first laboratory appointment will be an introductory training session which will comprise of collection of physiological eligibility measures (height, weight, waist-to-hip ratio, blood pressure) and training on the cognitive tasks, and sleep and wellbeing measures. Following this, the four testing visit appointments will be identical in procedure with the exception of the treatment administered.

For testing visits, participants will attend the research centre having abstained from alcohol (24 hours), over-the-counter medications (24 hours) and antihistamines (48 hours). There will be minimal restrictions to the participant in terms of abstinence from caffeine or food prior to testing visits; participants will be encouraged to follow their normal routine in regard to breakfast and caffeine consumption (whereby participants eat or do not eat breakfast based on what is usual for them). Participants must however consume their usual breakfast and caffeine no later than 1 hour prior to arrival and should ensure their breakfast and caffeine consumption is consistent across all 4 testing visits. Upon arrival, physiological measures will be collected including height and weight, blood pressure and waist-to-hip ratio. Participants will then complete a series of mood, wellbeing and sleep questionnaires including Visual Analogue Mood Scales (VAMS); Positive and Negative Affect Scale (PANAS); State Trait Anxiety Inventory (STAI); Depression, Anxiety and Stress Scale (DASS-21); Core Consensus Sleep Diary (CSD- Core); Sleep Quality Scale (SQS); World Health Organisation Quality of Life Questionnaire (WHOQOL-BREF). At testing visit 2 and 4 (Day 29 chronic visit, for each study arm) participants will complete the Caffeine Consumption Questionnaire to monitor changes to caffeine intake.

Following this, participants will complete a 50-minute computerised cognitive assessment administered via COMPASS including word, picture and face recognition, immediate word recall, delayed word recall, numeric working memory, choice reaction time, corsi blocks, peg and ball and cognitive demand battery (3 repetitions of serial 3 subtractions, serial 7 subtractions, rapid visual information processing task (RVIP) and 'mental fatigue' visual analogue scales).

After the COMPASS assessment, participants will consume their randomly allocated treatment for the day and a further blood pressure reading will be collected. An identical COMPASS assessment will be completed at 30 minutes post-dose. Following completion of the second COMPASS assessment, participants will be provided with their treatment to consume daily at home for the 29-day supplementation period. Participants will receive treatment consumption instructions and a treatment diary to write down the time treatment is taken each day. Participants will be instructed to return the completed treatment diary and all unused treatment at the following testing visit appointment (following the supplementation period).

For each study arm (each 29-day supplementation period) there will be 3 at home assessments for participants to complete via Qualtrics and Cognimapp. These will be a short series of sleep and wellbeing questionnaires, and a short battery of cognitive tasks, including VAMS, PANAS, SQS and Numeric Working Memory, Choice Reaction Time and Peg and Ball.

ELIGIBILITY:
Inclusion Criteria:

* You self-assess yourself as being in good health.
* You are aged 18-75 years at the time of giving consent.
* English is your first language or are fluent in English.

Exclusion Criteria:

* Insufficient (< 40 mg per day) or excessive (> 500 mg per day) habitual caffeine consumption (* NOTE: This will be calculated at screening but feel free to query this with the researcher prior to attendance.).
* Have any pre-existing medical conditions/illnesses which will impact taking part in the study. (* NOTE: The explicit exceptions to this are controlled hyper/hypothyroidism, hay fever, high cholesterol and reflux-related conditions. NOTE: There may be other, unforeseen, exceptions and these will be considered on a case-by-case basis, i.e. participants may be allowed to progress to screening if they have a condition/illness which would not interact with the active treatments or impede performance so it's worth discussing any medical conditions with the researcher prior to booking lab appointments).
* Are currently taking prescription medications which will impact taking part in the study (* NOTE: the explicit exceptions to this are contraceptive treatments for female participants, thyroid medications, topical skin treatments and those medications used in the treatment of high cholesterol and reflux-related conditions; and those taken 'as needed' in the treatment of asthma and hay fever.).
* Have high blood pressure (systolic over 139 mm Hg or diastolic over 89 mm Hg1) - *NOTE: We must measure this in the lab using our blood pressure monitors and can only use our measurements to access eligibility rather than home or GP readings.
* Have a Body Mass Index (BMI) outside of the range 18.5-39.9 kg/m2.
* Are pregnant, seeking to become pregnant or lactating.
* Have been diagnosed with a neurological condition or assessed as having a learning/behavioural or neurodevelopmental difference (e.g. dyslexia, autism, ADHD).
* Have a visual impairment that cannot be corrected with glasses or contact lenses (including colour-blindness).
* Smoke tobacco/ vape nicotine/ use nicotine replacement products (* NOTE: If participants have recently quit smoking or using replacements, they must have stopped using them altogether for a period of 3 months before participating in this study).
* Have relevant food allergies/ intolerances/ sensitivities (Please discuss all allergies/ intolerances/ sensitivities with the researcher prior to your screening appointment).
* Have taken antibiotics within the past 4 weeks.
* Are currently consuming any other dietary supplement (e.g., vitamins, omega 3 fish oils etc.) or have done so in the last 4 weeks. (* NOTE: Participation is possible following a 4-week supplement wash out prior to participating and for the duration of the study on the proviso that the supplements they are taking are out of choice and not medically prescribed or advised. Please discuss with the researcher if unsure. NOTE: We would never advise stopping supplements prescribed by your doctor e.g., iron, calcium etc., only those you use out of choice).
* Have any health conditions that would prevent the fulfilment of the study requirements (this includes non-diagnosed conditions for which no medication may be taken).
* Are unable to complete all of the study assessments (this will be assessed by the researcher at your training appointment, whereby you must be able to reach the minimum scores for each cognitive task to progress with the trial).
* Are currently participating in another clinical or nutrition intervention study or have done so in the past 4 weeks.
* Have been diagnosed with/ undergoing treatment for alcohol or drug abuse in the last 12 months.
* Have been diagnosed with/ undergoing treatment for a psychiatric disorder in the last 12 months, including a medical diagnosis of anxiety or depression.
* Suffer from frequent migraines that require medication (more than or equal to 1 per month).
* Have any sleep disorders or take any sleep aid medications.
* Have any known active infections.
* Will be non-compliant with regards to treatment consumption.
* Does not have a bank account (required for payment).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-02-24 (Estimated); Primary Completion 2025-12-19 (Estimated); Study Completion 2025-12-19 (Estimated)

PRIMARY OUTCOMES:
Attention - Cognitive domain factor score | Prior to (acute) and following 29-day chronic supplementation
  Effects of supplementation on the cognitive domain Attention, measured using the following tasks through the Computerised Mental Performance Assessment System (COMPASS, Northumbria University): Choice Reaction Time and Rapid Visual Information Processing. Scores of accuracies will be in the form of the percentage of responses correct and scores of performance speed will be reaction time measured in milliseconds, with lower scores indicating faster response time.

SECONDARY OUTCOMES:
Working Memory - Cognitive domain factor score | Prior to (acute) and following 29-day chronic supplementation
  Effects of supplementation on the cognitive domain Working Memory, measured using the following tasks through the Computerised Mental Performance Assessment System (COMPASS, Northumbria University): Numeric Working Memory (NWM), Serial 3s subtractions, Serial 7 subtractions and Corsi Blocks. Scores of accuracies will be in the form of the percentage of responses correct. For Numeric Working Memory task, scores of performance speed will be reaction time measured in milliseconds, with lower scores indicating faster response time.
Episodic Memory - Cognitive domain factor score | Prior to (acute) and following 29-day chronic supplementation
  Effects of supplementation on the cognitive domain Episodic Memory, measured using the following tasks through the Computerised Mental Performance Assessment System (COMPASS, Northumbria University): Immediate Word Recall, Delayed Word Recall, Delayed Name to Face Recall, Delayed Picture Recognition and Delayed Word Recognition. Scores of accuracies will be in the form of the percentage of responses correct. For the following tasks, scores of performance speed will be reaction time measured in milliseconds, with lower scores indicating faster response time: Delayed Name to Face Recall, Delayed Picture Recognition and Delayed Word Recognition.
Executive Function - Cognitive Domain factor score | Prior to (acute) and following 29-day chronic supplementation
  Effects of supplementation on the cognitive domain Executive Function, measured using the following tasks through the Computerised Mental Performance Assessment System (COMPASS, Northumbria University): Peg and Ball, and Cognitive Demand Battery (comprised of 3 repetitions of Serial 3s subtractions, Serial 7s subtractions and Rapid Visual Information Processing tasks). For Peg and Ball, scores will include average thinking time and completion time in milliseconds, with lower scores indicating faster response time, along with number of errors.
Choice Reaction Time | Days 7, 14 and 21, for both study arms
  Cognition task completed on smartphones via an online cognition website "Cognimapp" sent to participants via a link from the researcher at days 7, 14 and 21 of the supplementation periods. Performance on Choice Reaction Time task - accuracy and reaction time outcomes Cognitive task score, % and msecs.
Numeric Working Memory | Days 7, 14 and 21, for both study arms
  Cognition task completed on smartphones via an online cognition website "Cognimapp" sent to participants via a link from the researcher at days 7, 14 and 21 of the supplementation periods. Performance on Numeric Working Memory task - accuracy and reaction time outcomes Cognitive task score, % and msecs.
Peg and Ball | Days 7, 14 and 21, for both study arms
  Cognition task completed on smartphones via an online cognition website "Cognimapp" sent to participants via a link from the researcher at days 7, 14 and 21 of the supplementation periods. Performance on Peg and Ball task - average thinking time and completion time, msecs, and number of errors.
Self-Reported Mood via Visual Analogue Mood Scales (VAMS) | Prior to (acute) and following days 7, 14, 21 and 29 (chronic) of supplementation, for both study arms
  Subjective ratings of mood via digital Visual Analogue Mood Scales. 18 x 100mm lines anchored at either end by antonyms (e.g., 'alert-drowsy', 'calm-excited'). Outcomes - Scores from the VAMS can be collapsed into three measures, Alertness, Stress and Tranquillity.
Self-Reported Mood via Positive and Negative Affect Scale (PANAS) | Prior to (acute) and following days 7, 14, 21 and 29 (chronic) of supplementation, for both study arms
  Subjective ratings of positive and negative mood via Positive and Negative Affect Scale. 20 item measure, summed to create 2 component scores: negative affect (scores from 10-50) and positive affect (scores from 10-50). Items are answered on a 5-point Likert scale ranging from 1 (Very slightly or not at all) to 5 (Extremely). For the positive affect component, higher scores indicate higher levels of positive affect. For the negative affect component, lower scores indicate lower levels of negative affect.
Self-Reported Mood via Depression, Anxiety and Stress Scale (DASS-21) | Prior to (acute) and following 29-day chronic supplementation
  Subjective ratings of mood via Depression, Anxiety and Stress scale. 21 item measure, summed to create 3 component scores: depression (scores from 0-21), anxiety (scores from 0-21) and stress (scores from 0-21). Items are answered on a 4-point Likert scale ranging from 0 (Did not apply to me at all) to 3 (Applied to me very much or most of the time). An overall distress score can be calculated by summing the 3 component scores (scores from 0-63, with higher scores indicating higher overall distress). Higher component scores indicate higher depression, anxiety and stress.
Self-Reported Anxiety via State Trait Anxiety Inventory (STAI) | Prior to (acute) and following 29-day chronic supplementation
  Subjective ratings of anxiety via State Trait Anxiety Inventory. 40 item measure, summed to create 2 component scores: state anxiety (scores from 20-80) and trait anxiety (scores from 20-80). Items are answered on a 4-point Likert scale ranging from 1 (Almost never) to 4 (Almost always). Higher component scores indicate higher anxiety.
Self-Reported Wellbeing via World Health Organisation Quality of Life Scale (WHOQOL-BREF) | Prior to (acute) and following 29-day chronic supplementation
  Subjective ratings of wellbeing via World Health Organisation Quality of Life Scale. 26 item measure using a 5-point Likert scale to create 4 component scores: physical health (scores from 1-, psychological, social relationships and environment. Higher scores indicate higher quality of life. Scores for each component are created by calculating the average answer points for each domain and multiple the result by 4 (scores from 4-20). A total score can be calculated from the 4 component scores, ranging from 0-100, with higher scores indicating higher quality of life.
Self-Reported Sleep Quality via Sleep Quality Scale (SQS) | Prior to (acute) and following days 7, 14, 21 and 29 (chronic) of supplementation, for both study arms
  Subjective ratings of sleep quality via Sleep Quality Scale. 28 item measure encompassing 6 components: daytime symptoms, restoration after sleep, problems initiating sleep, problems maintaining sleep, difficulty waking and sleep satisfaction. Scores are summed to create a total score ranging between 0-84. Items are answered on a 4-point Likert scale ranging between 0 (Few) and 3 (Almost always). Higher scores indicate more acute sleep problems.
Self-Reported Sleep Continuity via Core Consensus Sleep Diary (CSD-Core) | Prior to (acute) and following 29-day chronic supplementation
  Subjective ratings of sleep continuity via Core Consensus Sleep Diary. 12 item measure utilised to calculate 7 components: sleep latency, time in bed, number of awakenings, wake after sleep onset, total sleep time, sleep efficiency and sleep quality. The sleep quality component is rated on a 4-point Likert scale ranging between 1 (Very poor) to 5 (Very good), with higher scores indicating higher sleep quality (total score from 0-5).
Systolic Blood Pressure | Prior to (acute) and following 29-day chronic supplementation
  Systolic blood pressure (mmHg)
Diastolic Blood Pressure | Prior to (acute) and following 29-day chronic supplementation
  Diastolic blood pressure (mmHg)
Heart Rate | Prior to (acute) and following 29-day chronic supplementation
  Hart rate (bpm)
Self-Reported Caffeine Consumption via Caffeine Consumption Questionnaire (CCQ) | Prior to (acute) and following 29-day chronic supplementation
  Subjective rating of caffeine consumption via Caffeine Consumption Questionnaire. Questionnaire containing 21 items used to measure self-reported daily intake, and the amount and type of caffeine product consumed (i.e., coffee, tea, energy drinks, chocolate). Higher scores indicates higher caffeine consumption.

CONTACTS AND LOCATIONS:
Locations (1):
- Brain Performance and Nutrition Research Centre- Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Immediately following publication with no end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose, such as for the purpose of a meta-analysis.
  Any named author on this project/publication will be able to approve and provide access to the IPD.